CLINICAL TRIAL: NCT06058949
Title: Health Protection and Promotion of Sign Language Interpreters Through Implementation of Total Worker Health®
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Gretchen Roman, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00008720; K01OH012441 (NIH)
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Well-Being, Psychological
Keywords: sign language interpreters; Total Worker Health®
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Protection and Promotion Program (Experimental)
  Interventions: Behavioral: Health Protection and Promotion
- General Health Program (Active Comparator)
  Interventions: Behavioral: General Health Program

INTERVENTIONS:
Behavioral: Health Protection and Promotion — An adaptive integrated Total Worker Health® program. Virtual 8-week program that's been contextualized to the physical and mental health needs of sign language interpreters. It will examine biomechanics, sleep hygiene, vicarious trauma and burnout, demand-control schema, physical activity, emotional management strategies, proper nutrition and examination of worksite.
  Arms: Health Protection and Promotion Program
Behavioral: General Health Program — Virtual 8-week program that addresses participant sleep hygiene, physical activity and proper nutrition.
  Arms: General Health Program

SUMMARY:
Using mixed-methods and a clinical efficacy trial design, the overall objective of this study will employ implementation strategies to adapt and evaluate a previous integrated Total Worker Health® (TWH®) program and pilot test its efficacy on sign language interpreter well-being. The central hypothesis is that interpreters in the health protection and promotion program (intervention) will demonstrate significantly improved well-being compared to those in a general health program (control).

ELIGIBILITY:
Inclusion Criteria:

* Bilingual in English and American Sign Language
* Certified sign language interpreter working at least 10 hours/week in any interpreter setting.
* Apparently healthy

Exclusion Criteria:

* Less than 18 year old
* Not yet certified as a sign language interpreter
* Unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
mean change in acceptability using the Training Acceptability Rating Scale-1 (TARS-1) | 15 to 24 months
  TARS-1 measures acceptability using six items (1=strongly disagree; 6=strongly agree) and demonstrates good test-retest reliability, internal consistency, and construct and concurrent validity. The scale ranges from 6 to 36 with higher scores indicating better acceptability.
mean change in acceptability using the Training Acceptability Rating Scale-2 (TARS-2) | 15 to 24 months
  TARS-2 assesses perceived impact with eight items (0=not at all; 3=a great deal) and demonstrates good face and concurrent validity. Of particular interest, TARS-2 also includes three qualitative items asking about the most helpful part of the program and any recommended changes and invites other comments. The scale ranges from 0-24 with higher scores indicating better outcomes.
mean change in Acceptability, Feasibility, and Appropriateness Scale | 15 to 24 months
  This acceptability (six items), feasibility (three items), and appropriateness (five items) instrument will be used to assess whether or not the intervention efforts were successful. The 14 total items across three subscales demonstrate good to excellent internal consistency and are rated on a five-point scale (1=not at all; 5=extremely). High scores of 30, 15, and 25 and low scores of 6, 3, and 5 indicate excellent and poor acceptability, feasibility, and appropriateness, respectively.
mean change in the National Institute of Occupational Safety and Health's Worker Well-Being Questionnaire- work evaluation and experience | baseline to post intervention (approximately 15-24 months)
  Work evaluation and experience is the first of five domains in this comprehensive measure of worker well-being and has 16 total questions. Total summed scores within this section range from 23-128 with higher scores indicating better outcomes (accounting for inverse scoring on negative items).
mean change in the National Institute of Occupational Safety and Health's Worker Well-Being Questionnaire- work evaluation and experience | baseline to 6 months post intervention (approximately 21-30 months)
  Work evaluation and experience is the first of five domains in this comprehensive measure of worker well-being and has 16 total questions. Total scores within this section range from 23-128 with higher scores indicating better outcomes (accounting for inverse scoring on negative items).
mean change in the National Institute of Occupational Safety and Health's Worker Well-Being Questionnaire- workplace policies and culture | baseline to post intervention (approximately 15-24 months)
  Workplace policies and culture is the second of five domains in this comprehensive measure of worker well-being and has 14 total questions. Total scores within this section range from 12-75 with higher scores indicating better outcomes (accounting for inverse scoring on negative items).
mean change in the National Institute of Occupational Safety and Health's Worker Well-Being Questionnaire- workplace policies and culture | baseline to 6 months post intervention (approximately 21-30 months)
  Workplace policies and culture is the second of five domains in this comprehensive measure of worker well-being and has 14 total questions. Total scores within this section range from 12-75 with higher scores indicating better outcomes (accounting for inverse scoring on negative items).
mean change in the National Institute of Occupational Safety and Health's Worker Well-Being Questionnaire- workplace physical environment and safety climate | baseline to post intervention (approximately 15-24 months)
  Workplace physical environment and safety climate is the third of five domains in this comprehensive measure of worker well-being and has 10 total questions. Total scores within this section range from 14-60 with higher scores indicating better outcomes (accounting for inverse scoring on negative items).
mean change in the National Institute of Occupational Safety and Health's Worker Well-Being Questionnaire- workplace physical environment and safety climate | baseline to 6 months post intervention (approximately 21-30 months)
  Workplace physical environment and safety climate is the third of five domains in this comprehensive measure of worker well-being and has 10 total questions. Total scores within this section range from 14-60 with higher scores indicating better outcomes (accounting for inverse scoring on negative items).
mean change in the National Institute of Occupational Safety and Health's Worker Well-Being Questionnaire- health status | baseline to post intervention (approximately 15-24 months)
  Health status is the fourth of five domains in this comprehensive measure of worker well-being and has 23 total questions. There are five open text box items within this section (i.e. asking for the number of days the respondent gets high intensity physical activity). Otherwise, total scores of the Likert scale items within this section range from 24-146 with higher scores indicating better outcomes (accounting for inverse scoring on negative items).
mean change in the National Institute of Occupational Safety and Health's Worker Well-Being Questionnaire- health status | baseline to 6 months post intervention (approximately 21-30 months)
  Health status is the fourth of five domains in this comprehensive measure of worker well-being and has 23 total questions. There are five open text box items within this section (i.e. asking for the number of days the respondent gets high intensity physical activity). Otherwise, total scores of the Likert scale items within this section range from 24-146 with higher scores indicating better outcomes (accounting for inverse scoring on negative items).
mean change in the National Institute of Occupational Safety and Health's Worker Well-Being Questionnaire- home, community, and society | baseline to post intervention (approximately 15-24 months)
  Home, community, and society is the final domain in this comprehensive measure of worker well-being and has 5 total questions. Total scores within this section range from 11-65 with higher scores indicating better outcomes (accounting for inverse scoring on negative items).
mean change in the National Institute of Occupational Safety and Health's Worker Well-Being Questionnaire- home, community, and society | baseline to 6 months post intervention (approximately 21-30 months)
  Home, community, and society is the final domain in this comprehensive measure of worker well-being and has 5 total questions. Total scores within this section range from 11-65 with higher scores indicating better outcomes (accounting for inverse scoring on negative items).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

REFERENCES:
- [Background] Eriksen HR, Ihlebaek C, Mikkelsen A, Gronningsaeter H, Sandal GM, Ursin H. Improving subjective health at the worksite: a randomized controlled trial of stress management training, physical exercise and an integrated health programme. Occup Med (Lond). 2002 Oct;52(7):383-91. doi: 10.1093/occmed/52.7.383. PMID 12422025
- [Background] Tveito TH, Eriksen HR. Integrated health programme: a workplace randomized controlled trial. J Adv Nurs. 2009 Jan;65(1):110-9. doi: 10.1111/j.1365-2648.2008.04846.x. Epub 2008 Nov 14. PMID 19032505